CLINICAL TRIAL: NCT03714139
Title: Immediate Loading-A Histological Study in Humans
Brief Title: Immediate Loading a Histological Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARDEC Academy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: dental implants
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Edentulous Alveolar Ridge
Keywords: Dental Implants; bone healing; clinical trial; histology
MeSH Terms: interventions — Immediate Dental Implant Loading; Prostheses and Implants

STUDY DESIGN:
Intervention Model Description: Split mouth, At least one site will be used as a test and one as a control where experimental mini-implants will be installed.
Who Masked: Investigator, Outcomes Assessor
Masking Description: One of the researchers , neither involved in the selection of the patients nor in the surgical and prosthetic treatment, will carry out electronically the randomization (randomization.com). Will be prepared sealed opaque envelopes and opened at the time of surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate implant Loading (Experimental): Immediate loading is defined as the placement of the implant and immediate prosthetic restoration
  Interventions: Procedure: immediate loading; Procedure: non implant loading
- non implant loading (No Intervention): there is not immediate prosthetic restoration

INTERVENTIONS:
Procedure: immediate loading — The participants will be assigned to immediate or delayed functional loading groups. In each participant, edentulous areas with adequate thickness of the alveolar bone crest will be identified and at least two sites will be identified for implant installation. All implant recipient sites will be sub-prepared to allow good stability of the implants. Experimental mini-implants (Sweden & Martina, Due Carrare, Padova, Italy), 3.5 mm in diameter and with an intraosseous portion of 4 mm in length will be installed.
  Immediate loading group - A prosthetic component will be applied over the trial implants. Impressions will be taken and a crown / bridge will be provided to patients in one day.
  Other Names: implant surgery, prosthesis
  Arms: Immediate implant Loading
Procedure: non implant loading — Control implants will receive a healing screw and will remain unloaded
  Other Names: control site
  Arms: Immediate implant Loading

SUMMARY:
Twelve participants with edentulous alveolar crests in the distal portion of the arches will be included in the study. At least two implant sites will be identified in each patient and will be sub-prepared with drills or sonic instruments. One site will be used as a test and one as a control where experimental mini-implants will be installed. Reconstructive surgical procedures will be applied at the biopsy sites.

DETAILED DESCRIPTION:
Objective: - To evaluate histologically the influence of the functional load on implants, both immediate and delayed.

Material and methods: 12 participants with edentulous alveolar crests in the distal portion of the arches will be included in the study. At least two implant sites will be identified in each patient and will be sub-prepared with drills or sonic instruments to obtain a high degree of torque to ensure optimum primary stability. At least one site will be used as a test and one as a control where experimental mini-implants will be installed. Test sites will be loaded immediately. The control sites will remain unloaded. After 2 months, mini-implants will be recovered as planned for each group. Reconstructive surgical procedures will be applied at the biopsy sites, if necessary, using autologous bone or bone substitutes and membranes. Standard implants will be installed during the same surgical session and, after 2 months, the planned prosthesis will be performed. Patients will be followed for at least 2 years for evaluation and intervention, if necessary.

Biopsies will be included in resin to obtain wear cuts for histomorphometric analysis. The bone histomorphometry will be evaluated and statistical analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥25 years of age) with the need of at least two implants to replace teeth of the jaw will be included.
* Natural antagonist teeth have to be present both at test and control sites to guarantee occlusal contacts

Exclusion Criteria:

* untreated rampant caries or uncontrolled periodontal disease of the remaining teeth
* diabetes not controlled diabetes or any other systemic or local disease that could compromise postoperative healing and / or osseointegration
* need for systemic corticosteroids or any other medication that could compromise postoperative healing and / or osseointegration
* inability or unwillingness to return to follow-up not likely to be able to comply with the study procedures according to the judgment of the investigators
* pregnancy

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — patients with edentulous spaces
Enrollment: 12 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
bone to implant contact | 2 months
  The linear distances between IS and B (IS-B) and CM and X (CM-X) were measured parallel to the long axis of the implant at both sides of the implant at a magnification of x100.
  Moreover, the amount of new bone, old bone, total bone (new + old bone = BIC%

SECONDARY OUTCOMES:
Bone density | 2 months
  The total amount of mineralized bone in contact with the implant surface measured histomorphometrically

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Botticelli, PHd, Study Director — ARDEC Academy
Locations (1):
- Colombia, Cartagena, Cartagena, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
there is a plan to save all the data to do the follow up

REFERENCES:
- [Background] Bousdras VA, Walboomers F, Jansen JA, Cunningham JL, Blunn G, Petrie A, Jaecques S, Naert IE, Sindet-Pedersen S, Goodship AE. Immediate functional loading of single-tooth TiO2 grit-blasted implant restoration. A controlled prospective study in a porcine model. Part II: Histology and histomorphometry. Clin Implant Dent Relat Res. 2007 Dec;9(4):207-16. doi: 10.1111/j.1708-8208.2007.00039.x. PMID 18031442
- [Background] Calandriello R, Tomatis M, Vallone R, Rangert B, Gottlow J. Immediate occlusal loading of single lower molars using Branemark System Wide-Platform TiUnite implants: an interim report of a prospective open-ended clinical multicenter study. Clin Implant Dent Relat Res. 2003;5 Suppl 1:74-80. doi: 10.1111/j.1708-8208.2003.tb00018.x. PMID 12691653
- [Background] Cecchinato D, Bressan EA, Toia M, Araujo MG, Liljenberg B, Lindhe J. Osseointegration in periodontitis susceptible individuals. Clin Oral Implants Res. 2012 Jan;23(1):1-4. doi: 10.1111/j.1600-0501.2011.02293.x. Epub 2011 Nov 1. PMID 22092689
- [Background] Degidi M, Petrone G, Lezzi G, Piattelli A. Histologic evaluation of 2 human immediately loaded and 1 titanium implants inserted in the posterior mandible and submerged retrieved after 6 months. J Oral Implantol. 2003;29(5):223-9. doi: 10.1563/1548-1336(2003)0292.3.CO;2. PMID 14620684
- [Background] Degidi M, Piattelli A, Shibli JA, Perrotti V, Iezzi G. Bone formation around immediately loaded and submerged dental implants with a modified sandblasted and acid-etched surface after 4 and 8 weeks: a human histologic and histomorphometric analysis. Int J Oral Maxillofac Implants. 2009 Sep-Oct;24(5):896-901. PMID 19865630
- [Background] Degidi M, Scarano A, Petrone G, Piattelli A. Histologic analysis of clinically retrieved immediately loaded titanium implants: a report of 11 cases. Clin Implant Dent Relat Res. 2003;5(2):89-93. doi: 10.1111/j.1708-8208.2003.tb00189.x. PMID 14536043
- [Result] Bosshardt DD, Salvi GE, Huynh-Ba G, Ivanovski S, Donos N, Lang NP. The role of bone debris in early healing adjacent to hydrophilic and hydrophobic implant surfaces in man. Clin Oral Implants Res. 2011 Apr;22(4):357-64. doi: 10.1111/j.1600-0501.2010.02107.x. PMID 21561477

DOCUMENTS (1):
  • Study Protocol (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT03714139/Prot_000.pdf